CLINICAL TRIAL: NCT05955235
Title: A Long-term Safety Follow-up Study of SCM-AGH in Patients Who Completed SCM-APT2001 Study
Status: Active, not recruiting | Type: Observational
Sponsor: SCM Lifescience Co., LTD. (Industry)
Responsible Party: Sponsor
Other Study IDs: APT2001-LTFU
Record Dates: First submitted 2023-06-23; First posted 2023-07-21 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-06

CONDITIONS: Pancreatitis, Acute
Keywords: Stem Cell Therapy; SCM-AGH; Pancreatitis
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Not Applicable(Observation Study) — Not Applicable(Observation Study)

SUMMARY:
This is a long-term safety follow-up study of the Phase I/IIa multicenter study of SCM-AGH in subjects with moderate to severe acute pancreatitis. subjects will be followed up for a maximum period of 240 weeks after the first dose of investigational product. Only subjects previously enrolled in protocol SCM-APT2001 (ClinicalTrials.gov ID: NCT04189419) will be eligible for this long-term follow-up protocol.

DETAILED DESCRIPTION:
Subjects who meet all eligibility criteria for Long Term Follow-Up(LTFU) study participation at the SCM-APT2001 End of Treatment(EOT) visit may continue LTFU for a maximum period of up to 240 weeks post first dose of investigational product. No additional dosing will be administered on this LTFU protocol.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who provide written informed consent
* Subjects who have received at least 1 dose of SCM-AGH in the SCM-APT2001 study

Exclusion Criteria:

* N/A

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects who have received at least 1 dose of SCM-AGH in the SCM-APT2001 study (ClinicalTrials.gov ID: NCT04189419)
Sampling Method: Non-Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2019-05-10 (Actual); Primary Completion 2026-08-20 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Long-term safety assessment | Up to 5 Years
  Ratio and number of cases for subjects who have experienced SAE(Serious Adverse Event).
Mortality | Up to 5 Years
  Ratio of subjects who died during long-term safety follow-up
Ratio of subjects with malignant tumors formed during the long-term safety follow-up period | Up to 5 Years
  The number, ratio, and number of cases of malignant tumor formation

SECONDARY OUTCOMES:
Number of occurrences of Abnormal, clinically significant in laboratory results | Up to 5 Years
  Perform if necessary.
  * Hematology: RBC, Hemoglobin, Hematocrit, Platelet count, WBC with Differential Count
  * Chemistry: Na, K, Ca, Cl, BUN, Creatinine, Uric acid, Total bilirubin, Albumin, Total protein, ALT, AST, r-GT, ALP, LDH, glucose, Total cholesterol, Triglyceride, C-reactive protein
  * Urinalysis: Protein, Glucose, Urobilinogen, WBC, RBC Blood coagulation test: aPTT, PT
Number of occurrences of Abnormal, clinically significant in Vital Signs | Up to 5 Years
  Measure systolic blood pressure, diastolic blood pressure, pulse, and body temperature.

CONTACTS AND LOCATIONS:
Locations (6):
- South Korea (6):
  - Soonchunhyang University Hosptial Bucheon, Bucheon-si, Gyenggi-do
  - Kyungpook National University Chilgok Hospital, Daegu
  - Dongguk University Ilsan Hospital, Goyang-si
  - Chonnam National University Medical School, Gwangju
  - Inha University Hospital, Incheon
  - Ajou University Hospital, Suwon